CLINICAL TRIAL: NCT00571649
Title: Multicenter, Randomized, Parallel-group Efficacy and Safety Study for the Prevention of Venous Thromboembolism in Hospitalized Medically Ill Patients Comparing Rivaroxaban With Enoxaparin. The MAGELLAN Study
Brief Title: Venous Thromboembolic Event (VTE) Prophylaxis in Medically Ill Patients
Acronym: MAGELLAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12839; 2007-004614-14 (EudraCT Number)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Venous Thromboembolism
Keywords: Acute medical illnesses with increased risk for VTE.; Deep vein thrombosis (DVT); Pulmonary embolism (PE),; Venous Thromboembolic disease (VTE),; Medical illness
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Xarelto, BAY59-7939) (Experimental): Participants received 10 mg oral rivaroxaban tablet once daily (OD) for 35 +/- 4 days, plus subcutaneous enoxaparin-matched placebo solution OD for 10 +/- 4 days
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939); Drug: Enoxaparin placebo
- Enoxaparin (Active Comparator): Participants received oral rivaroxaban-matched placebo tablet OD for 35 +/- 4 days, plus 40 mg subcutaneous enoxaparin solution OD for 10 +/- 4 days
  Interventions: Drug: Enoxaparin; Drug: Rivaroxaban placebo

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Oral rivaroxaban 10 mg once daily administered for 35 +/- 4 days
  Arms: Rivaroxaban (Xarelto, BAY59-7939)
Drug: Enoxaparin — Subcutaneous enoxaparin 40 mg once daily (OD) administered for 10 +/- 4 days
  Arms: Enoxaparin
Drug: Rivaroxaban placebo — Oral rivaroxaban-matched placebo tablet OD for 35 +/- 4 days
  Arms: Enoxaparin
Drug: Enoxaparin placebo — Subcutaneous enoxaparin-matched placebo solution OD for 10 +/- 4 days
  Arms: Rivaroxaban (Xarelto, BAY59-7939)

SUMMARY:
This study will evaluate if extended therapy with oral rivaroxaban can prevent blood clots in the leg and lung that can occur with patients hospitalized for acute medical illness, and compare these results with those of the standard enoxaparin dose and duration regimen. The safety of rivaroxaban will also be studied.

DETAILED DESCRIPTION:
The treatment period was followed by a follow-up period starting the day after the last intake of study medication, regardless of the actual duration of study drug administration and ended on Day 90 (+ 7 days). Participants who did not complete the treatment period also entered the follow-up period. It was also possible that participants did not enter the follow-up period, e.g. due to withdrawal of consent or termination of study participation.

Within the US 'Johnson & Johnson Pharmaceutical Research & Development, L.L.C.' is sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40 years or more
* Patients at risk of venous thromboembolic events being hospitalized for acute medical conditions as follows:

  * Heart failure, New York Heart Association (NYHA) class III or IV
  * Active cancer
  * Acute ischemic stroke
  * Acute infectious and inflammatory diseases, including acute rheumatic diseases
  * Acute respiratory insufficiency
  * Additional risk factor for VTE, including reduced mobility

Exclusion Criteria:

* Conditions that contraindicate the use of antithrombotic therapy with the Low Molecular-Weight Heparin (LMWH) enoxaparin
* Conditions that may increase the risk of bleeding, including intracranial hemorrhage
* Required drugs or procedures which may interfere with the study treatment
* Concomitant conditions or diseases which may increase the risk of study subjects or interfere with the study outcome
* General conditions in which subjects are not suitable to participate in the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8101 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (547):
- United States (110):
  - Birmingham, Alabama
  - Dothan, Alabama
  - Office of Dr. John Simmons, MD, Geneva, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Tuscaloosa, Alabama
  - Little Rock, Arkansas
  - Chula Vista, California
  - Duarte, California
  - Encinitas, California
  - Fountain Valley, California
  - Fullerton, California
  - Glendale, California
  - Oceanside, California
  - Pasadena, California
  - Redlands, California
  - Sacramento, California
  - San Diego, California
  - Santa Barbara, California
  - Torrance, California
  - Denver, Colorado
  - Pueblo, Colorado
  - Wheat Ridge, Colorado
  - Farmington, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Boyton Beach, Florida
  - Clearwater, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - Pembroke Pines, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Fort Gordon, Georgia
  - Savannah, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Springfield, Illinois
  - Anderson, Indiana
  - Noblesville, Indiana
  - Des Moines, Iowa
  - Olathe, Kansas
  - Lafayette, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Biddeford, Maine
  - Rockport, Maine
  - Baltimore, Maryland
  - Framingham, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Pontiac, Michigan
  - Saint Clair Shores, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Anaconda, Montana
  - Great Falls, Montana
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Somerville, New Jersey
  - Summit, New Jersey
  - Teaneck, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Jamaica, New York
  - New Hyde Park, New York
  - New York, New York
  - Stony Brook, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Elizabeth City, North Carolina
  - Greensboro, North Carolina
  - Fargo, North Dakota
  - Canton, Ohio
  - Columbus, Ohio
  - Maumee, Ohio
  - Toledo, Ohio
  - Bethlehem, Pennsylvania
  - Camp Hill, Pennsylvania
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Corsicana, Texas
  - Dallas, Texas
  - Edinburg, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Richmond, Virginia
  - Everett, Washington
  - Tacoma, Washington
  - Clarksburg, West Virginia
- Argentina (7):
  - Avellaneda, Buenos Aires
  - San Miguel, Buenos Aires
  - Hospital de Agudos "Dr. Carlos Bocalandro", Tres de Febrero, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Hospital Británico, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Sanatorio Mitre, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Vicente López
- Australia (15):
  - Garran, Australian Capital Territory
  - Kogarah, New South Wales
  - Lismore, New South Wales
  - Sydney, New South Wales
  - Auchenflower, Queensland
  - Brisbane, Queensland
  - Redcliffe, Queensland
  - Southport, Queensland
  - Woollongabba, Queensland
  - Adelaide, South Australia
  - Launceston, Tasmania
  - Box Hill, Victoria
  - Clayton, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Austria (15):
  - Kittsee, Burgenland
  - Oberpullendorf, Burgenland
  - Wolfsberg, Carinthia
  - Gratwein, Styria
  - Graz, Styria
  - Hartberg, Styria
  - Leoben, Styria
  - Zams, Tyrol
  - Linz, Upper Austria
  - Vienna, Vienna
  - Innsbruck
  - Linz
  - Mürzzuschlag
  - Sankt Pölten
  - Vienna
- Belgium (16):
  - Aalst
  - Bruges
  - Bruxelles - Brussel
  - Dendermonde
  - Hasselt
  - Huy
  - Ieper
  - Leuven
  - Malmedy
  - Mol
  - Montigny S/sambre
  - Mortsel
  - Roeselare
  - Sint-Niklaas
  - Tubize
  - Turnhout
- Brazil (5):
  - Curitiba, Paraná
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
- Bulgaria (6):
  - Pleven
  - Rousse
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo
- Canada (14):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Saint John, New Brunswick
  - Cobourg, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Hotel Dieu-Grace Hospital, Windsor, Ontario
  - Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Ste-Foy, Quebec
- Chile (2):
  - Santiago
  - Viña del Mar
- China (13):
  - Guangzhou, Guangdong
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Changchun, Jilin
  - Dalian, Liaoning
  - Shenyang, Liaoning
  - The 1st Affiliated Hosp of the 4th Military Med Uni, Xi'an, Shaanxi
  - 1st Affiliated Hosp., Med College Xi'an Jiaotong Univ., Xi'an, Shaanxi
  - Chengdu, Sichuan
  - Beijing
  - Beijing Friendship Hosp., Beijing
  - Chongqing
  - Shanghai
- Colombia (6):
  - Medellín, Antioquia
  - Bogotá, Bogota D.C.
  - Cali, Valle del Cauca Department
  - Bogotá
  - Cali
  - Medellín
- Croatia (4):
  - Osijek
  - Rijeka
  - Zadar
  - Zagreb
- Czechia (8):
  - Brno
  - Kutná Hora
  - Nové Město na Moravě
  - Olomouc
  - Pilsen
  - Prague
  - Říčany
  - Znojmo
- Denmark (6):
  - Esbjerg
  - Frederiksberg C
  - Kolding
  - København NV
  - København S
  - Roskilde
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (7):
  - Hämeenlinna
  - Helsinki
  - Jyväskylä
  - Lahti
  - Lappeenranta
  - Raisio
  - Turku
- France (24):
  - Arras
  - Besançon
  - Brest
  - Castelnau-le-Lez
  - Clermont-Ferrand
  - Colombes
  - Dijon
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Montpellier
  - Nice
  - Nîmes
  - Paris
  - Pierre-Bénite
  - Reims
  - Roubaix
  - Saint-Etienne
  - Saint-Herblain
  - Strasbourg
  - Toulouse
  - Tourcoing
  - Vandœuvre-lès-Nancy
- Germany (28):
  - Bad Mergentheim, Baden-Wurttemberg
  - Esslingen am Neckar, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsbad, Baden-Wurttemberg
  - Weiden, Bavaria
  - Beeskow, Brandenburg
  - Frankfurt (Oder), Brandenburg
  - Bremen, City state Bremen
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Jülich, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Neuss, North Rhine-Westphalia
  - Oberhausen, North Rhine-Westphalia
  - Paderborn, North Rhine-Westphalia
  - Soest, North Rhine-Westphalia
  - Stolberg, North Rhine-Westphalia
  - Troisdorf, North Rhine-Westphalia
  - Viersen, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Neuwied, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Pirna, Saxony
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin
- Greece (7):
  - Elefsina, Attica
  - Kifisia / Athens, Attica
  - Abelokipi - Athens
  - Athens
  - Nea Ionia
  - Piraeus
  - Rio / Patras
- Hong Kong (2):
  - Shatin, N.t.
  - Shatin
- Hungary (10):
  - Baja
  - Balassagyarmat
  - Budapest
  - Debrecen
  - Győr
  - Hódmezővásárhely
  - Kecskemét
  - Székesfehérvár
  - Tatabánya
  - Zalaegerszeg-Pozva
- India (12):
  - Ahmedabad, Gujar?t
  - Bangalore, Karn?taka
  - Calicut, Kerala
  - Thiruvananthapuram, Kerala
  - Pune, Maharashtra
  - Ludhiana, Punjab
  - Chennai, Tamil N?du
  - Coimbatore, Tamil N?du
  - Kolkata, West Bengal
  - Hyderabad
  - Mumbai
  - Noida
- Indonesia (2):
  - Jakarta
  - Surabaya
- Israel (8):
  - Afula
  - Ashkelon
  - Haifa
  - Holon
  - Kfar Saba
  - Rehovot
  - Safed
  - Tel Aviv
- Italy (21):
  - Acquaviva delle Fonti, Bari
  - Napoli, Campania
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Varese, Lombardy
  - Campobasso, Molise
  - Fidenza, Parma
  - Catania, Sicily
  - Palermo, Sicily
  - Terni, Trentino-Alto Adige
  - Perugia, Umbria
  - Domodossola, Verbano-Cusio-Ossola
  - Bergamo
  - Latina
  - Reggio Calabria
  - Vicenza
- Japan (33):
  - Ichinomiya, Aichi-ken
  - Kasugai, Aichi-ken
  - Ōbu, Aichi-ken
  - Matsuyama, Ehime
  - Tōon, Ehime
  - Fukui-shi, Fukui
  - Chikushino-shi, Fukuoka
  - Takasaki, Gunma
  - Kure, Hiroshima
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Amagasaki, Hyōgo
  - National Hospital Organization Ibaraki Higashi Hospital, Ibaraki, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Hanamaki, Iwate
  - Ebina, Kanagawa
  - Kamakura, Kanagawa
  - Yokohama, Kanagawa
  - Nangoku, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Matsusaka, Mie-ken
  - Tsu, Mie-ken
  - Kashiwazaki, Niigata
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Daitō, Osaka
  - Yao, Osaka
  - Kusatsu, Shiga
  - Hamamatsu, Shizuoka
  - Meguro-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Shimonoseki, Yamaguchi
- Latvia (5):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
  - Ventspils
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Utena
  - Vilnius
- Luxembourg (3):
  - Luxembourg
  - Luxembourg-Kirchberg
  - Niedercorn
- Malaysia (3):
  - Kuala Lumpur
  - Negeri Sembilan,
  - Sarawak
- Mexico (16):
  - Aguascalientes, Aguascalientes
  - Tuxtla Gutiérrez, Chiapas
  - Chihuahua City, Chihuahua
  - Torreón, Coahuila
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Mexico D. F., Mexico City
  - México, D.F, Mexico City
  - México, D.F., Mexico City
  - Morelia, Michoacán
  - Monterrey, Nuevo León
  - Puebla City, Puebla
  - Hermosillo, Sonora
  - Metepec, State of Mexico
  - Mérida, Yucatán
  - Zacatecas City, Zacatecas
- Netherlands (9):
  - Amersfoort
  - Amsterdam
  - Enschede
  - Heerlen
  - Maastricht
  - Nieuwegein
  - Rotterdam
  - Sittard
  - Utrecht
- New Zealand (2):
  - Auckland
  - Christchurch
- Norway (4):
  - Fredrikstad
  - Gjøvik
  - Hamar
  - Oslo
- Pakistan (2):
  - Karachi
  - Lahore
- Peru (3):
  - Callao
  - Lima
  - Lima Cercado
- Poland (12):
  - Bialystok
  - Bydgoszcz
  - Krakow
  - Lublin
  - Olsztyn
  - Piotrkow Trybunalski
  - Siedlce
  - Starogard Gdański
  - Szczecin
  - Tarnów
  - Warsaw
  - Włocławek
- Portugal (11):
  - S. Martinho Do Bispo, Coimbra District
  - Lisbon, Lisbon District
  - Porto, Porto District
  - Santarém, Santarém District
  - Amadora
  - Cascais
  - Coimbra
  - Lisbon
  - Matosinhos Municipality
  - Porto
  - Viana do Castelo
- Romania (3):
  - Bucharest
  - Constanța
  - Suceava
- Russia (3):
  - Moscow
  - Nizhny Novgorod
  - Yaroslavl
- Singapore (2):
  - Singapore
  - Changi General Hospital, Singapore
- Slovakia (4):
  - Bratislava
  - Lučenec
  - Martin
  - Žilina
- Slovenia (3):
  - Golnik
  - Ljubljana
  - Novo Mesto
- South Africa (10):
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Pretoria, Gauteng
  - Roodepoort, Gauteng
  - Sandton, Gauteng, South Africa
  - Goodwood, Western Cape
  - Somerset West, Western Cape
  - Stellenbosch, Western Cape
  - Worcester, Western Cape
- South Korea (6):
  - Gyeongi-do, Korea
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Seoul Metropolitan Boramae Hospital, Seoul, Seoul Teugbyeolsi
  - Gyeonggi-do
  - Jeollanam-do
  - Seoul
- Spain (12):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Sabadell, Barcelona
  - Cuenca, Cuenca
  - Cabra, Córdoba
  - Córdoba, Córdoba
  - Girona, Girona
  - Olot, Girona
  - Cartagena, Murcia
  - Vélez, Málaga
  - Vigo, Pontevedra
  - Zaragoza, Zaragoza
- Sweden (11):
  - Borås
  - Hässleholm
  - Karlshamn
  - Kristianstad
  - Lund
  - Malmo
  - Skövde
  - Stockholm
  - Sundsvall
  - Umeå
  - Visby
- Switzerland (9):
  - Bruderholz, Basel-Landschaft
  - Basel, Canton of Basel-City
  - Liestal, Canton of Basel-City
  - Bern, Canton of Bern
  - Langenthal, Canton of Bern
  - Geneva, Canton of Geneva
  - Zurich, Canton of Zurich
  - Baden
  - Lucerne
- Taiwan (3):
  - Kaohsiung City
  - Tainan
  - Taipei
- Thailand (3):
  - Bangkok, Thailand
  - Bangkok
  - Chiang Mai
- Turkey (Türkiye) (2):
  - Istanbul
  - Izmir
- Ukraine (8):
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Simferopol
- United Kingdom (10):
  - Middlesbrough, Cleveland
  - Dumfries, Dumfries and Galloway
  - London, London
  - Liverpool, Merseyside
  - Sheffield, South Yorkshire
  - Glasgow, Stratchclyde
  - Newcastle upon Tyne, Tyne and Wear
  - Leeds, West Yorkshire
  - London
  - Nottingham

REFERENCES:
- [Result] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos A, Tapson V. Extended-duration rivaroxaban thromboprophylaxis in acutely ill medical patients: MAGELLAN study protocol. J Thromb Thrombolysis. 2011 May;31(4):407-16. doi: 10.1007/s11239-011-0549-x. PMID 21359646
- [Result] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos AC, Tapson V; MAGELLAN Investigators. Rivaroxaban for thromboprophylaxis in acutely ill medical patients. N Engl J Med. 2013 Feb 7;368(6):513-23. doi: 10.1056/NEJMoa1111096. PMID 23388003
- [Result] Sharma A, Chatterjee S, Lichstein E, Mukherjee D. Extended thromboprophylaxis for medically ill patients with decreased mobility: does it improve outcomes? J Thromb Haemost. 2012 Oct;10(10):2053-60. doi: 10.1111/j.1538-7836.2012.04874.x. PMID 22863355
- [Result] Mebazaa A, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Merli G, Schellong SW, Spyropoulos AC, Tapson VF, De Sanctis Y, Cohen AT. Predicting the risk of venous thromboembolism in patients hospitalized with heart failure. Circulation. 2014 Jul 29;130(5):410-8. doi: 10.1161/CIRCULATIONAHA.113.003126. Epub 2014 Jun 26. PMID 24970782
- [Result] Cohen AT, Spiro TE, Spyropoulos AC, Desanctis YH, Homering M, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Tapson VF, Burton P; MAGELLAN Study Group. D-dimer as a predictor of venous thromboembolism in acutely ill, hospitalized patients: a subanalysis of the randomized controlled MAGELLAN trial. J Thromb Haemost. 2014 Apr;12(4):479-87. doi: 10.1111/jth.12515. PMID 24460645
- [Derived] Spyropoulos AC, Raskob GE, Cohen AT, Ageno W, Weitz JI, Spiro TE, Lu W, Lipardi C, Albers GW, Elliott CG, Halperin JL, Hiatt WR, Maynard G, Steg PG, Sugarmann C, Barnathan ES. Association of Bleeding Severity With Mortality in Extended Thromboprophylaxis of Medically Ill Patients in the MAGELLAN and MARINER Trials. Circulation. 2022 May 10;145(19):1471-1479. doi: 10.1161/CIRCULATIONAHA.121.057847. Epub 2022 Apr 7. PMID 35389229
- [Derived] Raskob GE, Spyropoulos AC, Spiro TE, Lu W, Yuan Z, Levitan B, Suh E, Barnathan ES. Benefit-Risk of Rivaroxaban for Extended Thromboprophylaxis After Hospitalization for Medical Illness: Pooled Analysis From MAGELLAN and MARINER. J Am Heart Assoc. 2021 Nov 16;10(22):e021579. doi: 10.1161/JAHA.121.021579. Epub 2021 Nov 10. PMID 34755519
- [Derived] Raskob GE, Spyropoulos AC, Cohen AT, Weitz JI, Ageno W, De Sanctis Y, Lu W, Xu J, Albanese J, Sugarmann C, Weber T, Lipardi C, Spiro TE, Barnathan ES. Association Between Asymptomatic Proximal Deep Vein Thrombosis and Mortality in Acutely Ill Medical Patients. J Am Heart Assoc. 2021 Feb;10(5):e019459. doi: 10.1161/JAHA.120.019459. Epub 2021 Feb 15. PMID 33586478
- [Derived] Jamil A, Jamil U, Singh K, Khan F, Chi G. Extended Thromboprophylaxis With Betrixaban or Rivaroxaban for Acutely Ill Hospitalized Medical Patients: Meta-Analysis of Prespecified Subgroups. Crit Pathw Cardiol. 2021 Mar 1;20(1):16-24. doi: 10.1097/HPC.0000000000000232. PMID 32657973
- [Derived] Weitz JI, Raskob GE, Spyropoulos AC, Spiro TE, De Sanctis Y, Xu J, Lu W, Suh E, Argenti D, Yang H, Albanese J, Lipardi C, Barnathan ES. Thromboprophylaxis with Rivaroxaban in Acutely Ill Medical Patients with Renal Impairment: Insights from the MAGELLAN and MARINER Trials. Thromb Haemost. 2020 Mar;120(3):515-524. doi: 10.1055/s-0039-1701009. Epub 2020 Jan 23. PMID 31975354
- [Derived] Chi G, Goldhaber SZ, Kittelson JM, Turpie AGG, Hernandez AF, Hull RD, Gold A, Curnutte JT, Cohen AT, Harrington RA, Gibson CM. Effect of extended-duration thromboprophylaxis on venous thromboembolism and major bleeding among acutely ill hospitalized medical patients: a bivariate analysis. J Thromb Haemost. 2017 Oct;15(10):1913-1922. doi: 10.1111/jth.13783. Epub 2017 Sep 4. PMID 28762617
- [Derived] Marszalek J, Mehrsefat S, Chi G. The risk of stroke among acutely ill hospitalized medical patients: lessons from recent trials on extended-duration thromboprophylaxis. Expert Rev Hematol. 2017 Aug;10(8):679-684. doi: 10.1080/17474086.2017.1343662. Epub 2017 Jun 21. PMID 28617144
- See also: Click here and search for results of Bayer Products provided by EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit date: 04 DEC 2007; last patient last visit date 24 NOV 2010. Primary completion date: 12 AUG 2010. Participants were aged ≥40 years, hospitalized for an acute medical illness, and at risk of Venous Thromboembolism (VTE) (with heart failure, cancer, ischemic stroke, infection or inflammation, or respiratory insufficiency)
Pre-assignment Details: A total of 8428 participants were screened; 327 failed. 8101 were randomized. 7998 (98.7%) were in the Safety Analysis Set (SAF), i.e. received study medication. 6024 (74.4%) were in the modified Intent to Treat (at Day 35) group (valid for SAF with adequate assessment of venous thromboembolism). A total of 6005 (74.1%) completed study.
Groups:
- Rivaroxaban (Xarelto, BAY59-7939): Participants received 10 mg oral rivaroxaban tablet once daily (OD) for 35 +/- 4 days, plus subcutaneous enoxaparin-matched placebo solution OD for 10 +/- 4 days during treatment period
- Enoxaparin: Participants received oral rivaroxaban-matched placebo tablet OD for 35 +/- 4 days, plus 40 mg subcutaneous enoxaparin solution OD for 10 +/- 4 days during treatment period
Period: Treatment Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Started | 4050 | 4051
Participants Received Treatment | 3997 | 4001
Day 10 | 3454 | 3499
Day 35 | 3033 | 3115
Completed | 2958 | 3047
Not Completed | 1092 | 1004
Not completed — Adverse Event | 438 | 385
Not completed — Clinical endpoint reached | 50 | 56
Not completed — Withdrawal by Subject | 285 | 255
Not completed — Death | 76 | 59
Not completed — Physician Decision | 8 | 9
Not completed — Lost to Follow-up | 43 | 41
Not completed — Non-compliant with study medication | 88 | 89
Not completed — Patient convenience | 11 | 13
Not completed — Protocol Violation | 90 | 92
Not completed — Technical problems | 3 | 5
Period: Follow-up Period
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Started | 3583 (Participants were required to enter follow-up even if treatment period not completed.) | 3635 (Participants were required to enter follow-up even if treatment period not completed.)
Completed | 3038 (Began day after last dose study drug; ended on Day 90 (+/- 7 days) .) | 3107 (Began day after last dose study drug; ended on Day 90 (+/- 7 days) .)
Not Completed | 545 | 528
Not completed — Adverse Event | 46 | 40
Not completed — Clinical endpoint reached | 5 | 2
Not completed — Withdrawal by Subject | 119 | 115
Not completed — Death | 132 | 133
Not completed — Physician Decision | 7 | 13
Not completed — Lost to Follow-up | 95 | 92
Not completed — Patient convenience | 136 | 121
Not completed — Protocol Violation | 5 | 12

BASELINE CHARACTERISTICS:
Groups:
- Rivaroxaban (Xarelto, BAY59-7939): Participants received 10 mg oral rivaroxaban tablet once daily (OD) for 35 +/- 4 days, plus subcutaneous enoxaparin-matched placebo solution OD for 10 +/- 4 days (SAF population)
- Enoxaparin: Participants received oral rivaroxaban-matched placebo tablet OD for 35 +/- 4 days, plus 40 mg subcutaneous enoxaparin solution OD for 10 +/- 4 days (SAF population)
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin | Total
Number analyzed (Participants) | 3997 | 4001 | 7998
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (11.9) | 69.2 (11.7) | 69.2 (11.8)
Age, Customized [Number; unit: participants]
  < 65 years | 1323 | 1363 | 2686
  65 to < 75 years | 1144 | 1090 | 2234
  >= 75 years | 1530 | 1548 | 3078
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1774 | 1898 | 3672
  Male | 2223 | 2103 | 4326
Race [Number; unit: participants]
  White | 2749 | 2744 | 5493
  Black | 89 | 92 | 181
  Asian | 793 | 794 | 1587
  Native American | 12 | 12 | 24
  Hispanic | 69 | 70 | 139
  Uncodable | 106 | 112 | 218
  Unknown | 1 | 0 | 1
  Missing | 178 | 177 | 355
Reason for hospitalization [Number; unit: participants] — Participants may have more than one acute condition as hospitalization reason. Acute medical illnesses included heart failure (New York Heart Association [NYHA] Class III [marked limitation of physical activity] or NYHA Class IV [inability to carry out any physical activity without discomfort)] active cancer, acute ischemic stroke, acute infectious and inflammatory diseases (including acute rheumatic diseases), acute respiratory insufficiency.
  participants
    Heart failure (NYHA Class III or NYHA Class IV) | 1292 | 1301 | 2593
    Active cancer | 294 | 290 | 584
    Acute ischemic stroke | 691 | 692 | 1383
    Acute Infectious and Inflammatory Diseases | 1904 | 1876 | 3780
    Acute infectious disease | 1826 | 1801 | 3627
    Acute inflammatory or rheumatic disease | 150 | 149 | 299
    Acute respiratory insufficiency | 1085 | 1151 | 2236

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Endpoint of Venous Thromboembolism [VTE] (Any Deep Vein Thrombosis [DVT], Non Fatal Pulmonary Embolism [PE]) and VTE-related Death up to Day 35 + 6 Days
Description: A composite endpoint of: asymptomatic proximal DVT in lower extremity detected by mandatory bilateral lower extremity venous ultrasonography; symptomatic DVT in lower extremity, proximal or distal; symptomatic, non-fatal PE; and VTE-related death.
Time Frame: Up to Day 35 + 6 days
Population: modified Intent-to-Treat (mITT) Day 35: participant was valid for the safety analysis and had an adequate assessment of VTE up to Day 35
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 2967 | 3057
Percentage of participants | 4.4 | 5.7
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; A sample size of 2876 valid patients per group was estimated to obtain a joint power of at least 90% for both primary endpoints (91.4% for superiority) with 4% event rate at day 35 for comparator and 40% relative risk reduction; Test type: Superiority or Other; p = 0.0211, Cochran-Mantel-Haenszel — Hochberg procedure: A 2-sided p-value of less than 0.05 would be considered significant, if the 1-sided p-value of the other primary efficacy outcome measure was less than 0.025, elsewise a p-value of less than 0.025 would be considered significant; Weighted relative risks were calculated using asymptotic methods, with weights based upon sample sizes per strata (geographic region); Risk Ratio (RR) = 0.771, 95% CI [0.618 to 0.962]

2. Primary Outcome: Percentage of Participants With Composite Endpoint of VTE (Any DVT, Non Fatal PE) and VTE-related Death up to Day 10 + 5 Days
Description: as for outcome 1
Time Frame: Up to Day 10 + 5 days
Population: Per Protocol (PP) Day 10: participant was valid for the safety analysis, had an adequate assessment of VTE up to Day 10 not later than 48 hours after stop of study drug, met inclusion criteria, and had no major protocol deviations.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 2938 | 2993
Percentage of participants | 2.7 | 2.7
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; A sample size of 2876 valid patients per group was estimated to obtain a joint power of at least 90% for both primary endpoints (98.6% power for non-inferiority) with 1.8% event rate at day 10 for comparator and 35% relative risk reduction; Test type: Non-Inferiority or Equivalence — Rivaroxaban would be considered at least as effective as the comparator if the upper limit of the CI (Confidence Interval) was less than 1.5; p = 0.0025, Cochran-Mantel-Haenszel — Hochberg procedure: A 1-sided p-value of less than 0.025 would be considered significant, if the 2-sided p-value of the other primary efficacy outcome measure was less than 0.05, elsewise a p-value of less than 0.0125 would be considered significant; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.968, 95% CI [0.713 to 1.314]

3. Secondary Outcome: Percentage of Participants With Composite Endpoint of VTE (Any DVT, Non Fatal PE) and All-cause Mortality up to Day 35 + 6 Days
Description: A composite endpoint of: asymptomatic proximal DVT in lower extremity detected by mandatory bilateral lower extremity venous ultrasonography; symptomatic DVT in lower extremity, proximal or distal; symptomatic, non-fatal PE; and death (VTE-related and not VTE-related).
Time Frame: Up to Day 35 + 6 days
Population: modified Intent-to-Treat (mITT) Day 35 (participant was valid for the safety analysis and had an adequate assessment of VTE up to Day 35) expanded to include participants who had an assessment of all deaths, including not VTE-related
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3096 | 3169
Percentage of participants | 8.6 | 9.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; Test type: Superiority or Other; p = 0.3758, Cochran-Mantel-Haenszel — Test hierarchy: A p-value of less than 0.05 would be considered significant, if the tests for the two primary efficacy outcome measures were significant; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.931, 95% CI [0.795 to 1.091]

4. Secondary Outcome: Percentage of Participants With Composite Endpoint of VTE (Any DVT, Non Fatal PE) and VTE-related Death up to Day 10 + 5 Days Per mITT Population
Description: as for outcome 1
Time Frame: Up to Day 10 + 5 days
Population: modified Intent-to-Treat (mITT) Day 10: participant was valid for the safety analysis and had an adequate assessment of VTE up to Day 10
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3232 | 3271
Percentage of participants | 3.0 | 3.1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; Test type: Superiority or Other; p = 0.9473, Cochran-Mantel-Haenszel — Test hierarchy: A p-value of less than 0.05 would be considered significant, if the tests for the 2 primary efficacy outcomes and for "Composite endpoint of VTE (any DVT, non fatal PE) and all-cause mortality up to Day 35 + 6 days" were significant; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.991, 95% CI [0.753 to 1.304]

5. Secondary Outcome: Percentage of Participants With VTE Combined With All-cause Mortality up to Day 10 + 5 Days
Description: as for outcome 3
Time Frame: Up to Day 10 + 5 days
Population: modified Intent-to-Treat (mITT) Day 10 (participant was valid for the safety analysis and had an adequate assessment of VTE up to Day 10) expanded to include participants who had an assessment of all deaths, including not VTE-related
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3281 | 3310
Percentage of participants | 4.8 | 4.5

6. Secondary Outcome: Percentage of Participants With Symptomatic VTE, Including and Excluding VTE-related Death up to Days 10, 35, and 90
Description: Symptomatic VTE (non-fatal PE and DVT in lower extremity), including and excluding VTE-related death (PE and PE cannot be excluded) up to Days 10, 35, and 90
Time Frame: At Day 10 + 5 days, at Day 35 + 6 days, and at Day 90 + 7 days
Population: Safety population: Participant had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3997 | 4001
Percentage of participants
  symptomatic VTE (incl. VTE-related death)-Day 10 | 0.7 | 0.6
  symptomatic VTE (non fatal)-Day 10 | 0.5 | 0.3
  symptomatic VTE (incl. VTE-related death)-Day 35 | 1.0 | 1.4
  symptomatic VTE (non fatal)-Day 35 | 0.6 | 0.7
  symptomatic VTE (incl. VTE-related death)-Day 90 | 1.7 | 1.9
  symptomatic VTE (non fatal)-Day 90 | 0.7 | 0.9

7. Secondary Outcome: Percentage of Participants With Net Clinical Benefit (Any DVT, Non-fatal PE, VTE-related Death, Plus Major and Clinically Relevant Non-major Bleeding Events) up to Day 35 + 6 Days
Description: Net clinical benefit is a composite of the primary efficacy endpoint (asymptomatic proximal DVT in lower extremity detected by mandatory bilateral lower extremity venous ultrasonography; symptomatic DVT in lower extremity, proximal or distal; symptomatic, non-fatal PE; and VTE-related death) plus major and clinically relevant non-major bleeding events.
Time Frame: Up to Day 35 + 6 days
Population: modified Intent-to-Treat (mITT) Day 35 (participant was valid for the safety analysis and had an adequate assessment of VTE up to Day 35) expanded to include participants with major and clinically relevant bleeding events.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3042 | 3082
Percentage of participants | 9.4 | 7.8

8. Secondary Outcome: Percentage of Participants With Net Clinical Benefit (Any DVT, Non-fatal PE, VTE-related Death, Plus Major and Clinically Relevant Non-major Bleeding Events) up to Day 10 + 5 Days
Description: as for outcome 7
Time Frame: Up to Day 10 + 5 days
Population: Participants valid for safety analysis, with adequate assessment of VTE (to Day 10 within 48 hours of study drug), met inclusion criteria, and no major protocol deviations; expanded to include participants who had major bleeding or clinically relevant non-major bleeding events and met all criteria for PP except valid assessment of thromboembolism.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 2950 | 3007
Percentage of participants | 4.5 | 3.9

9. Secondary Outcome: Percentage of Participants With Major Vascular Events up to Days 10, 35, and 90
Description: Major vascular events included cardiovascular death, acute myocardial infarction (MI), or acute ischemic stroke. Participants may have had a vascular event in more than one category.
Time Frame: At Day 10 + 5 days, at Day 35 + 6 days, and at Day 90 + 7 days
Population: Safety population: Participant had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3997 | 4001
Percentage of participants
  Any event-Day 10 | 1.0 | 1.0
  Ischemic stroke-Day 10 | 0.3 | 0.3
  Acute MI-Day 10 | 0.5 | 0.4
  Death (cardiovascular)-Day 10 | 0.4 | 0.4
  Any event-Day 35 | 1.8 | 1.6
  Ischemic stroke-Day 35 | 0.5 | 0.5
  Acute MI-Day 35 | 0.6 | 0.5
  Death (cardiovascular)-Day 35 | 0.9 | 0.8
  Any event-Day 90 | 2.8 | 2.8
  Ischemic stroke-Day 90 | 0.8 | 1.1
  Acute MI-Day 90 | 0.9 | 0.7
  Death (cardiovascular)-Day 90 | 1.4 | 1.4

10. Secondary Outcome: Percentage of Participants With Each Component of the Composite Endpoint of VTE (Any DVT, Non Fatal PE) and VTE-related Death up to Day 35 + 6 Days
Description: The components of the composite endpoint include asymptomatic proximal DVT in lower extremity detected by mandatory bilateral lower extremity venous ultrasonography; symptomatic DVT in lower extremity, proximal or distal; symptomatic, non-fatal PE; and VTE-related death.
Time Frame: Up to Day 35 + 6 days
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 2967 | 3057
Percentage of participants
  Symptomatic non-fatal PE | 0.3 | 0.5
  Symptomatic DVT in lower extremity | 0.4 | 0.5
  Asymptomatic proximal DVT in lower extremity | 3.5 | 4.4
  VTE related death | 0.6 | 1.0

11. Secondary Outcome: Percentage of Participants With Each Component of the Composite Endpoint of VTE (Any DVT, Non Fatal PE) and VTE-related Death up to Day 10 + 5 Days
Description: as for outcome 10
Time Frame: Up to Day 10 + 5 days
Population: Per Protocol Day 10: participant was valid for the safety analysis, had an adequate assessment of VTE up to Day 10 not later than 48 hours after stop of study drug, met inclusion criteria, and had no major protocol deviations
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 2938 | 2993
Percentage of participants
  Symptomatic non-fatal PE | 0.2 | 0.1
  Symptomatic DVT in lower extremity | 0.2 | 0.2
  Asymptomatic proximal DVT in lower extremity | 2.4 | 2.4
  VTE related death | 0.1 | 0.2

12. Secondary Outcome: Percentage of Participants With All-cause Mortality up to Day 90 + 7 Days
Description: All deaths, including VTE-related deaths, cardiovascular deaths, and other deaths.
Time Frame: Up to Day 90 + 7 days
Population: Safety population: Participant had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3997 | 4001
Percentage of participants
  Any event | 6.7 | 6.2
  Death (cardiovascular) | 1.4 | 1.4
  Death (other) | 4.3 | 3.7
  VTE related death | 1.0 | 1.1

13. Secondary Outcome: Percentage of Participants With the Composite of Treatment Emergent Major Bleeding Events and Non-major Clinically Relevant Bleeding Events up to 2 Days After Last Intake of Any Study Medication (Day 35 + 6 Days)
Description: Major bleeding events were defined as events leading to >=2 g/dL fall in hemoglobin; or transfusion of >= 2 units of packed RBCs (Red blood cells) or whole blood; or leading to death. Non-major bleeding events were defined as overt bleeding not meeting the criteria of major bleeding
Time Frame: Up to Day 35 + 6 days
Population: Safety population: Participant had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3997 | 4001
Percentage of participants | 4.1 | 1.7
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; There was no sample size estimation as this was not planed as confirmatory analysis; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — 2-sided p-value. No adjustment for multiple testing; [statistical method as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.455, 95% CI 2-sided [1.854 to 3.251]

14. Secondary Outcome: Percentage of Participants With the Composite of Treatment Emergent Major Bleeding Events and Non-major Clinically Relevant Bleeding Events up to 2 Days After Last Application of a Study Medication Syringe (Day 10 + 5 Days)
Description: Major bleeding events were defined as events leading to >=2 g/dL fall in hemoglobin or transfusion of >=2 units of packed RBCs or whole blood or leading to death. Non-major bleeding events were defined as overt bleeding not meeting the criteria of major bleeding.
Time Frame: Up to Day 10 + 5 days
Population: Safety population: Participant had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Number analyzed (Participants) | 3997 | 4001
Percentage of participants | 2.8 | 1.2
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) vs Enoxaparin; There was no sample size estimation as this was not planed as confirmatory analysis; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — 2-sided p-value. No adjustment for multiple testing; Risk Ratio (RR) = 2.272, 95% CI 2-sided [1.628 to 3.171]

ADVERSE EVENTS:
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 1034/3997 | 976/4001
Other Adverse Events (participants affected / at risk) | 2297/3997 | 2291/4001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=3997) | Enoxaparin (N=4001)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 18 (20) | 13 (13)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13) | 9 (9)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 30 (31) | 28 (29)
Angina pectoris (Cardiac disorders) | 1 (1) | 4 (4)
Angina unstable (Cardiac disorders) | 6 (7) | 6 (6)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 6 (6)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 23 (23) | 22 (24)
Atrial flutter (Cardiac disorders) | 5 (5) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 5 (5)
Bradycardia (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac arrest (Cardiac disorders) | 12 (13) | 11 (12)
Cardiac failure (Cardiac disorders) | 76 (84) | 76 (81)
Cardiac failure acute (Cardiac disorders) | 11 (12) | 25 (28)
Cardiac failure chronic (Cardiac disorders) | 10 (10) | 10 (11)
Cardiac failure congestive (Cardiac disorders) | 31 (37) | 31 (38)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 11 (11) | 12 (12)
Cardiogenic shock (Cardiac disorders) | 6 (6) | 4 (4)
Cardiomegaly (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (2)
Cor pulmonale (Cardiac disorders) | 1 (1) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 2 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 12 (13) | 7 (8)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 3 (3) | 6 (6)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 3 (3)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 4 (6) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 7 (8) | 1 (2)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 3 (3)
Atrial thrombosis (Cardiac disorders) | 4 (4) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Electromechanical dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 5 (5) | 8 (8)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Haemorrhage coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Rheumatic heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Myotonic dystrophy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0)
Pupils unequal (Eye disorders) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Entropion (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 10 (11)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 (12) | 7 (8)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 3 (3)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 6 (6) | 3 (3)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (7)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 4 (5)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (5)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 4 (4) | 1 (1)
Chest pain (General disorders) | 10 (10) | 16 (18)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 14 (14) | 9 (9)
Fatigue (General disorders) | 2 (2) | 3 (3)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 8 (8) | 5 (5)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 5 (6)
Pain (General disorders) | 4 (4) | 2 (3)
Pyrexia (General disorders) | 8 (8) | 9 (9)
Sudden death (General disorders) | 8 (8) | 5 (5)
Performance status decreased (General disorders) | 0 (0) | 2 (3)
Hernia pain (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) | 7 (7)
General physical health deterioration (General disorders) | 5 (5) | 4 (4)
Puncture site haemorrhage (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 1 (1)
Unevaluable event (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Implant site haematoma (General disorders) | 0 (0) | 1 (1)
Device malfunction (General disorders) | 0 (0) | 1 (1)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0)
Disuse syndrome (General disorders) | 0 (0) | 1 (1)
Device capturing issue (General disorders) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 3 (4)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 4 (4)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Granulomatous liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 7 (7) | 5 (5)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Acquired immunodeficiency syndrome (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchiectasis (Infections and infestations) | 3 (3) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 18 (18) | 4 (4)
Bronchopneumonia (Infections and infestations) | 8 (8) | 10 (10)
Cellulitis (Infections and infestations) | 20 (23) | 9 (10)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 5 (5) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 2 (3)
Enteritis necroticans (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 4 (4) | 2 (2)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 12 (12) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 2 (2)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Lung abscess (Infections and infestations) | 2 (2) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 4 (4) | 1 (1)
Peridiverticular abscess (Infections and infestations) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 74 (78) | 76 (78)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2)
Pyometra (Infections and infestations) | 0 (0) | 1 (1)
Pyothorax (Infections and infestations) | 1 (1) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 29 (30) | 14 (14)
Septic shock (Infections and infestations) | 15 (16) | 18 (20)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 17 (20) | 13 (14)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 6 (6)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Burn infection (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis syndrome (Infections and infestations) | 1 (1) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 10 (10) | 12 (12)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 3 (3) | 0 (0)
Wound sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis liver (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 2 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 4 (4)
Pneumonia fungal (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 10 (12) | 6 (6)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye penetration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple drug overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 20 (20) | 23 (26)
Arteriogram coronary (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (7)
Biopsy lymph gland (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (4) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (2) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 4 (4) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (3) | 1 (1)
Immunoglobulins increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 8 (8) | 5 (5)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0)
Aspiration bronchial (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 3 (3) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 10 (10) | 11 (11)
Occult blood positive (Investigations) | 1 (1) | 2 (2)
Coagulation test (Investigations) | 1 (1) | 0 (0)
False positive investigation result (Investigations) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 4 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Diabetic foot (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 4 (4)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
Colorectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Ovarian epithelial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloma recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (18) | 11 (11)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 2 (2)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral circulatory failure (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 3 (3) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 2 (2) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 3 (3)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 2 (2)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 3 (3) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 3 (3) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 4 (4) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 15 (18) | 10 (10)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 10 (10)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1)
Quadriparesis (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 2 (2) | 3 (3)
Vascular dementia (Nervous system disorders) | 1 (1) | 2 (2)
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 30 (31) | 39 (40)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Critical illness polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute polyneuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 3 (3) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 5 (5)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 2 (2) | 1 (1)
Somatisation disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 1 (2)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (2)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (2)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (9) | 7 (7)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 12 (12) | 14 (14)
Renal failure acute (Renal and urinary disorders) | 31 (32) | 16 (16)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis glandularis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
Pulmonary renal syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Penile haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 35 (37) | 12 (13)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 109 (138) | 104 (131)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 17 (18)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 10 (11)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (12)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 14 (14)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 56 (59) | 40 (41)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Disability (Social circumstances) | 1 (1) | 0 (0)
Social problem (Social circumstances) | 1 (1) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Radical hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral artery angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Tumour excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Chemotherapy (Surgical and medical procedures) | 2 (2) | 2 (2)
Mitral valve repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 3 (5) | 3 (3)
Aortic thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial rupture (Vascular disorders) | 1 (2) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 2 (2)
Arteriosclerosis (Vascular disorders) | 3 (3) | 0 (0)
Arteritis (Vascular disorders) | 1 (1) | 1 (1)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 2 (2)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 4 (4)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 10 (10) | 7 (7)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 2 (2)
Iliac artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 3 (3) | 5 (5)
Shock (Vascular disorders) | 2 (2) | 3 (3)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 5 (5)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Superior vena caval occlusion (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (3) | 2 (2)
Arteriosclerosis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection rupture (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) (N=3997) | Enoxaparin (N=4001)
Anaemia (Blood and lymphatic system disorders) | 87 (93) | 85 (87)
Neutropenia (Blood and lymphatic system disorders) | 20 (32) | 16 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (32) | 25 (27)
Atrial fibrillation (Cardiac disorders) | 74 (82) | 61 (65)
Cardiac failure (Cardiac disorders) | 43 (46) | 38 (44)
Mitral valve incompetence (Cardiac disorders) | 36 (36) | 32 (33)
Tachycardia (Cardiac disorders) | 32 (33) | 43 (49)
Tricuspid valve incompetence (Cardiac disorders) | 19 (19) | 22 (22)
Ventricular extrasystoles (Cardiac disorders) | 24 (26) | 17 (17)
Vertigo (Ear and labyrinth disorders) | 26 (26) | 25 (26)
Conjunctivitis (Eye disorders) | 16 (16) | 24 (24)
Abdominal pain (Gastrointestinal disorders) | 89 (109) | 56 (64)
Abdominal pain upper (Gastrointestinal disorders) | 59 (63) | 53 (62)
Constipation (Gastrointestinal disorders) | 362 (418) | 346 (375)
Diarrhoea (Gastrointestinal disorders) | 214 (238) | 230 (256)
Dyspepsia (Gastrointestinal disorders) | 53 (54) | 62 (69)
Gastritis (Gastrointestinal disorders) | 36 (37) | 38 (38)
Gastritis erosive (Gastrointestinal disorders) | 20 (21) | 19 (19)
Gingival bleeding (Gastrointestinal disorders) | 20 (22) | 9 (9)
Hiatus hernia (Gastrointestinal disorders) | 20 (20) | 16 (16)
Nausea (Gastrointestinal disorders) | 207 (242) | 226 (253)
Vomiting (Gastrointestinal disorders) | 170 (205) | 149 (175)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 22 (23) | 12 (12)
Asthenia (General disorders) | 52 (54) | 31 (32)
Chest pain (General disorders) | 89 (102) | 77 (82)
Fatigue (General disorders) | 33 (35) | 35 (35)
Injection site haemorrhage (General disorders) | 8 (8) | 21 (23)
Oedema peripheral (General disorders) | 132 (153) | 115 (127)
Pain (General disorders) | 42 (46) | 39 (40)
Pyrexia (General disorders) | 132 (158) | 131 (162)
Cholelithiasis (Hepatobiliary disorders) | 49 (50) | 47 (48)
Hepatic function abnormal (Hepatobiliary disorders) | 17 (18) | 24 (24)
Hepatic steatosis (Hepatobiliary disorders) | 48 (48) | 61 (61)
Bronchitis (Infections and infestations) | 64 (65) | 47 (48)
Cellulitis (Infections and infestations) | 22 (22) | 18 (19)
Nasopharyngitis (Infections and infestations) | 37 (38) | 36 (36)
Oral candidiasis (Infections and infestations) | 31 (31) | 34 (35)
Pneumonia (Infections and infestations) | 73 (75) | 65 (68)
Upper respiratory tract infection (Infections and infestations) | 30 (33) | 26 (27)
Urinary tract infection (Infections and infestations) | 138 (148) | 142 (151)
Fall (Injury, poisoning and procedural complications) | 33 (38) | 40 (40)
Contusion (Injury, poisoning and procedural complications) | 38 (50) | 42 (63)
Alanine aminotransferase increased (Investigations) | 32 (32) | 61 (66)
Aspartate aminotransferase increased (Investigations) | 23 (23) | 35 (36)
Blood creatinine increased (Investigations) | 38 (40) | 36 (39)
Blood urea increased (Investigations) | 24 (27) | 23 (24)
Creatinine renal clearance decreased (Investigations) | 36 (40) | 35 (35)
Gamma-glutamyltransferase increased (Investigations) | 31 (31) | 32 (32)
Haemoglobin decreased (Investigations) | 23 (26) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 43 (49) | 30 (30)
Diabetes mellitus (Metabolism and nutrition disorders) | 39 (40) | 34 (34)
Hyperglycaemia (Metabolism and nutrition disorders) | 46 (54) | 50 (63)
Hyperkalaemia (Metabolism and nutrition disorders) | 62 (66) | 51 (57)
Hypoglycaemia (Metabolism and nutrition disorders) | 37 (46) | 39 (48)
Hypokalaemia (Metabolism and nutrition disorders) | 191 (219) | 184 (219)
Hyponatraemia (Metabolism and nutrition disorders) | 35 (38) | 34 (34)
Decreased appetite (Metabolism and nutrition disorders) | 38 (42) | 40 (44)
Arthralgia (Musculoskeletal and connective tissue disorders) | 62 (68) | 76 (87)
Back pain (Musculoskeletal and connective tissue disorders) | 97 (105) | 82 (85)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 (25) | 28 (30)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 46 (50) | 61 (66)
Neck pain (Musculoskeletal and connective tissue disorders) | 14 (14) | 22 (25)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29 (30) | 22 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 110 (127) | 103 (113)
Dizziness (Nervous system disorders) | 81 (83) | 72 (80)
Headache (Nervous system disorders) | 205 (237) | 185 (221)
Syncope (Nervous system disorders) | 23 (24) | 19 (21)
Anxiety (Psychiatric disorders) | 89 (99) | 94 (98)
Confusional state (Psychiatric disorders) | 28 (28) | 23 (24)
Depression (Psychiatric disorders) | 68 (68) | 73 (77)
Insomnia (Psychiatric disorders) | 172 (199) | 185 (202)
Sleep disorder (Psychiatric disorders) | 25 (25) | 16 (18)
Dysuria (Renal and urinary disorders) | 22 (23) | 15 (15)
Haematuria (Renal and urinary disorders) | 65 (68) | 48 (53)
Renal cyst (Renal and urinary disorders) | 65 (65) | 61 (63)
Renal failure (Renal and urinary disorders) | 52 (55) | 47 (48)
Renal failure acute (Renal and urinary disorders) | 25 (26) | 19 (19)
Urinary retention (Renal and urinary disorders) | 22 (23) | 17 (19)
Renal impairment (Renal and urinary disorders) | 39 (40) | 29 (31)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 44 (45) | 20 (20)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 71 (92) | 59 (84)
Cough (Respiratory, thoracic and mediastinal disorders) | 107 (118) | 94 (100)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 107 (120) | 99 (112)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 123 (145) | 66 (83)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 37 (40) | 32 (37)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 28 (32) | 31 (32)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 27 (28)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 21 (22) | 18 (23)
Ecchymosis (Skin and subcutaneous tissue disorders) | 42 (47) | 39 (42)
Erythema (Skin and subcutaneous tissue disorders) | 27 (30) | 37 (41)
Pruritus (Skin and subcutaneous tissue disorders) | 47 (47) | 50 (51)
Rash (Skin and subcutaneous tissue disorders) | 41 (44) | 50 (51)
Haematoma (Vascular disorders) | 24 (29) | 24 (26)
Hypertension (Vascular disorders) | 154 (177) | 156 (178)
Hypertensive crisis (Vascular disorders) | 20 (23) | 16 (18)
Hypotension (Vascular disorders) | 82 (91) | 93 (102)
Phlebitis (Vascular disorders) | 37 (38) | 38 (41)
Aortic arteriosclerosis (Vascular disorders) | 25 (25) | 19 (19)

LIMITATIONS AND CAVEATS:
A heterogeneous population (with different acute medical illnesses and severity of illness) was included in the trial. VTE risk in acute medical illnesses is moderate [with no thromboprophylaxis] .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days